CLINICAL TRIAL: NCT07011914
Title: CARE in MS: Childhood Adversity Research Effort in MS
Brief Title: Care in Multiple Sclerosis (MS)
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24-00939; 1R01NS139999 (NIH)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aim 1: Adults with RRMS - Focus Groups: Aim 1 will involve 2-3 focus groups, each with 8-12 participants per group. The focus group sessions will occur only one time and will take around 90-120 minutes. Aim 1 will enroll individuals with RRMS who self-identify as a Black, Hispanic, or poverty-impacted.
- Aim 2: Young Adults with MS - MRI Scan: Participants enrolled in Aim 2 will complete a baseline visit and research MRI occurring around and in concurrence with their routine/standard of care visit. The study visit is estimated to take around 1 to 1.5 hours. The MRI scan is estimated to take 30 minutes. The research team will maintain contact with study participants at least annually (up to 4 years).
  Aim 2 will enroll 330 young adults, of whom 165 have pediatric-onset RRMS and 165 have adult-onset RRMS. Further, 70% of participants in Aim 2 must self-identify as persons with MS who are either Black, Hispanic, or poverty-impacted.
- Aim 3: Young Adults with MS - Interviews: Aim 3 will involve one-time interviews estimated to take 30 to 45 minutes to complete. Aim 3 will enroll 20 participants who have completed at least 80% of study data in Aim 2; further, 70% of participants enrolled Aim 3 participants must self-identify as Black, Hispanic, or meet criteria for poverty impacted.

SUMMARY:
This study is structured around three main aims.

In Aim 1, investigators will conduct community-based participatory research (CBPR) to develop culturally tailored methods to assess childhood adversity in multiple sclerosis (MS).

Aim 2 will investigate the impact of childhood adversity on MS outcomes among individuals with relapsing-remitting MS (RRMS), among whom 70% belong to a group historically under-represented in MS research: Black, Hispanic, or poverty-impacted. Aim 2 procedures involve two visits that include a research blood draw and an MRI scan.

In Aim 3, investigators will conduct interviews and surveys to explore environmental and social factors affecting quality of life for minority MS patients.

ELIGIBILITY:
Inclusion Criteria:

Aim 1 -

* aged ≥18-29 years
* diagnosis of RRMS (Fulfill international criteria for relapsing remitting (RRMS))
* 70% self-identifying as a Black, Hispanic, or poverty-impacted (up to 138% of the federal poverty level) individual,and
* fluent in English or Spanish.

Aim 2 -

* aged ≥18-29 years
* diagnosis of RRMS (Fulfill international criteria for relapsing remitting (RRMS))
* 70% self-identifying as a Black, Hispanic, or poverty impacted, and
* fluent reading in English or Spanish
* Pediatric onset MS (MS onset before age 18 and age at time of enrollment is 18-25) OR adult-onset MS (MS onset at age 18 or older and age at time of enrollment is 19-29)
* Disease duration below 8 years

Aim 3 -

Aim 3 will enroll the first 20 participants from Aim 2 who meet the following criteria:

* completed at least 80% of study data in the cross-sectional study/Aim 2.
* a total of 70% must self-identify as Black, Hispanic, or meet criteria for poverty impacted.
* interviews will be evenly split between participants with high (top quartile) and low (bottom quartile) of PROMIS-10 scores.

Exclusion Criteria:

* Primary or Secondary Progressive MS
* Inability to consent.
* MS relapse within 30 days prior to study entry
* Other major neurologic or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Aim 1: 2-3 focus groups, each with 8-12 participants per group., aged ≥18 years with RRMS, who self-identify as a Black, Hispanic, or poverty-impacted, and are fluent in English or Spanish.
  * Aim 2: 330 young adults (ages 18-29 years of age with MS duration of 8 years or less) of whom 165 have pediatric-onset RRMS (aged 18-25) and 165 have adult-onset (aged 19-29) RRMS. 70% self-identify as persons with MS who are either Black, Hispanic, or poverty-impacted.
  * Aim 3: 20 participants who have completed at least 80% of study data in the cross-sectional study/Aim 2. 70% must self-identify as Black, Hispanic, or meet criteria for poverty impacted.
Sampling Method: Non-Probability Sample
Enrollment: 386 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Severity of MS | Baseline
  Severity of MS will be measured by MRI FLAIR lesion volume among Aim 2 participants.

SECONDARY OUTCOMES:
Age of MS Onset | Baseline
  Age of MS onset will be measured by interval between date of birth and MS symptom onset.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Krupp, MD, Principal Investigator — NYU Langone Health
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: kimberly.oneill@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to kimberly.oneill@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.